CLINICAL TRIAL: NCT00671125
Title: A Phase III, Randomized, Double-Blind Placebo-Controlled, PSG Plus Outpatient Study to Determine the Safety and Efficacy of TAK-375 in Adults With Chronic Insomnia
Brief Title: Study of Efficacy of Ramelteon in Adults With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-021; U1111-1114-8329 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Insomnia
Keywords: Sleep Disorder; Insomnia; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 16 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once nightly for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Ramelteon — Ramelteon 16 mg, tablets, orally, once nightly for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 16 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once nightly for up to 5 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Ramelteon, once daily (QD), in the treatment of chronic insomnia using polysomnography and subjective measures of sleep

DETAILED DESCRIPTION:
Insomnia is characterized by difficulties initiating and maintaining sleep or of nonrestorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a selective melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

This study will determine the safety and efficacy of 35-day treatment of chronic insomnia with Ramelteon using polysomnography and subjective measures of sleep. Participation in this study is anticipated to be about 2 months.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Females who are not of childbearing potential must be postmenopausal for 1 year or have history of hysterectomy and/or oophorectomy.
* Primary insomnia as defined by the DSM-IV-TRTM for at least 3 months and as defined by subjective sleep latency (sSL) greater than or equal to 30 minutes, subjective total sleep time (sTST) less than or equal to 6.5 hours per night, and daytime complaint(s) associated with disturbed sleep.
* Mean latency of greater than or equal to 20 minutes on 2 consecutive screening nights with neither night less than 15 minutes. Also, a mean of 60 minutes of wake time during the 480 minutes in bed across two nights with no night less than 45 minutes screening nights with neither night less than 15 minutes. Also, a mean of 60 minutes of wake time during the 480 minutes in bed across two nights with no night less than 45 minutes.
* Habitual bedtime is between 8:30 p.m. and 12:00 a.m.
* Body mass index between 18 and 34, inclusive.

Exclusion Criteria

* Known hypersensitivity to Ramelteon or related compounds, including melatonin.
* Previously participated in a study involving Ramelteon.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first night single-blind study medication, whichever is longer.
* Sleep schedule changes required by employment (e.g. shift worker) within three months prior to the first night of single-blind study medication, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the first night of single blind study medication.
* Ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes 4 or more alcoholic drinks per day.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to the first night of single-blind study medication.
* Uses tobacco products during nightly awakenings.
* Used melatonin, or other drugs or supplements known to affect sleep/wake function within 1 week (or 5 half lives of the drug, whichever is longer) prior to the first day of single-blind study medication.
* Used any central nervous system medication within 1 week (or 5 half lives of the drug, whichever is longer) prior to the first day of single-blind study medication. These medications must not have been used to treat psychiatric disorders.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Positive urine drug screen including alcohol at screening or a positive breathalyzer test at each check-in.
* Apnea hypopnea index (per hour of sleep) greater than 10 as seen on polysomnogram, on the first night of the polysomnogram screening.
* Periodic leg movement with arousal index (per hour of sleep) greater than 10 as seen on polysomnogram, on the first night of polysomnogram screening.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep/wake function
  * prohibit the subject from completing the study
  * not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Hypnotics
  * Antidepressants
  * Anticonvulsants
  * Sedating H1 antihistamines
  * Systemic steroids
  * Respiratory stimulants (eg, theophylline)
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Over-the-counter and prescription diet aids
  * Central nervous system active drugs (including herbal preparations with central nervous system effects)
  * Narcotic analgesics
  * All beta blockers
  * Melatonin
  * St. John's Wort
  * Kavakava
  * Gingko biloba

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 405 (Actual)
Dates: Start 2003-01; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Mean Latency to Persistent Sleep. | Week 1

SECONDARY OUTCOMES:
Mean Latency to Persistent Sleep. | Weeks 3 and 5 or Final Visit
Total Sleep Time. | Weeks 1, 3 and 5 or Final Visit
Sleep Efficiency. | Weeks 1, 3 and 5 or Final Visit
Awake Time after Persistent Sleep. | Weeks 1, 3 and 5 or Final Visit
Number of Awakenings after Persistent Sleep. | Weeks 1, 3 and 5 or Final Visit
Subjective Sleep Latency. | Weeks 1, 3 and 5 or Final Visit
Subjective Total Sleep Time. | Weeks 1, 3 and 5 or Final Visit
Subjective Sleep Quality. | Weeks 1, 3 and 5 or Final Visit
Subjective Awake Time. | Weeks 1, 3 and 5 or Final Visit
Subjective Number of Awakenings. | Weeks 1, 3 and 5 or Final Visit
Subjective Ease of Falling Back to Sleep. | Weeks 1, 3 and 5 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (25):
- United States (25):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Hot Springs, Arkansas
  - Anaheim, California
  - Oakland, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Miami, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Overland Park, Kansas
  - Crestview Hills, Kentucky
  - Chevy Chase, Maryland
  - Newton, Massachusetts
  - Troy, Michigan
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - New York, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Lafayette Hill, Pennsylvania
  - Austin, Texas
  - Plano, Texas

REFERENCES:
- [Result] Zammit G, Erman M, Wang-Weigand S, Sainati S, Zhang J, Roth T. Evaluation of the efficacy and safety of ramelteon in subjects with chronic insomnia. J Clin Sleep Med. 2007 Aug 15;3(5):495-504. PMID 17803013
- [Result] Mini L, Wang-Weigand S, Zhang J. Ramelteon 8 mg/d versus placebo in patients with chronic insomnia: post hoc analysis of a 5-week trial using 50% or greater reduction in latency to persistent sleep as a measure of treatment effect. Clin Ther. 2008 Jul;30(7):1316-23. doi: 10.1016/s0149-2918(08)80056-2. PMID 18691991
- [Result] Osborne, T, Louis, M, Wang-Weigand, S and Jie, Z. Treatment of insomnia in women and the melatonin receptor agonist ramelteon (Rozerem). Women's Health Care: A Practical Journal for Nurse Practitioners. 2008; 7: (6): 24-30
- [Result] Wang-Weigand S, McCue M, Ogrinc F, Mini L. Effects of ramelteon 8 mg on objective sleep latency in adults with chronic insomnia on nights 1 and 2: pooled analysis. Curr Med Res Opin. 2009 May;25(5):1209-13. doi: 10.1185/03007990902858527. PMID 19327100
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI